CLINICAL TRIAL: NCT00455260
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study, to Assess Tolerability, Safety, Pharmacokinetic and Pharmacodynamic Profiles of hGH-ViaDerm™ System in Adult Subjects With Growth Hormone Deficiency
Brief Title: A Multi-Dose Study to Assess Tolerability, Safety and Pharmacology of hGH-ViaDerm™ System in Adults With GH-Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry); TransPharma Medical (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GH-VD-102
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2009-04

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hGH-ViaDerm™ System (hGH or somatropin) — transdermal patch; Group 1: 0.2 mg/day SC hGH during Period I, and 0.5 mg per transdermal patch during Period III (expected equivalent dose to SC 0.2 mg/day) Group 2: 0.4 mg/day SC hGH during Period I, and 2.0 mg per transdermal patch during Period III (expected equivalent dose to SC 0.4 mg/day) Group 3: 1.0 mg/day SC hGH during Period I, and 5.0 mg per transdermal patch during Period III (expected equivalent dose to 1.0 mg/day)
Device: hGH-ViaDerm™ System — The hGH-ViaDerm™ System is a transdermal delivery system for somatropin (hGH, rDNA origin).
  The ViaDerm System™ consists of a medical device component and a printed dry hGH patch component. The device component is comprised of two primary elements: a reusable, computer mouse-like electronic controller and a disposable sterile array, which is inserted onto the base of the controller, delivers RF-current to ablate cells and creates microscopic throughways, termed RF-MicroChannels™, across the stratum corneum into the upper epidermis. The drug component consists of a unique circular transdermal dry hGH patch formulated specifically for use with the ViaDerm™ device. hGH is delivered by passive diffusion through the RF-MicroChannels™ into the systemic circulation system.

SUMMARY:
This study aims to examine the safety, tolerability and pharmacokinetics of transdermal delivery of human Growth Hormone (hGH or somatropin) using the ViaDerm device in adult patients with Growth Hormone Deficiency Syndrome.

ELIGIBILITY:
Inclusion Criteria:

Ages Eligible for Study: 20 Years - 60 Years, Genders Eligible for Study: Both

1. Clinical diagnosis of Adult Growth Hormone Deficiency (AGHD) meeting one of the following criteria:

   * Three or more additional pituitary hormone deficiencies, based on well documented medical history from up to 10 years prior to screening, and/or serum IGF-1 levels below 2 SD from normal level, measured up to 4 months prior to screening.
   * One or two additional pituitary hormone deficiencies with one GH stimulating test performed within 10 years prior to screening: Insulin Tolerance test with GH levels less than 5.1 µg/L or ARG-GHRH with GH levels less than 4.1 µg/L.
   * Isolated GH deficient subjects with two well-documented GH stimulating tests performed within 10 years prior to screening. Insulin Tolerance test with GH levels less than 5.1 µg/L or ARG-GHRH with GH levels less than 4.1 µg/L.
   * In childhood onset AGHD, confirmation of GHD following attainment of full height.
2. Subjects using hormone replacement therapy for additional pituitary deficits must be on an optimized treatment regimen for at least three months prior to screening.
3. Willing and able to provide written informed consent prior to performing any study procedures.

Exclusion Criteria:

1. GH therapy within one month prior to study entry.
2. For female subjects: pregnancy or lactation or use of oral contraception or unacceptable method of contraception throughout the study.
3. Active acromegaly in the last 5 years.
4. Carpal tunnel syndrome.
5. Prader-Willi syndrome.
6. Active Cushing's syndrome within the last 12 months.
7. Non-compliance for upper arm SC injection or patch application.
8. Skin color or tattoo that would not enable detection of erythema.
9. Upper extremities with skin marks, bruises, cuts, abrasions on the upper arm.
10. Dense and dark hair growth on upper extremities.
11. History of skin hypersensitivity and/or allergies.
12. Known hypersensitivity to somatropin or mannitol
13. Evidence of active malignancy.
14. Previous use of chemotherapy, immunosuppressive or radiation therapy, except for treatment of pituitary disease.
15. Serum glucose (fasting) > 126 mg/dl.
16. Known or suspected HIV-positive subjects or subjects with advanced diseases such as AIDS, Hepatitis C, Hepatitis B or tuberculosis.
17. Subjects who, based on the investigator's judgment, have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may include cardiovascular, vascular, pulmonary, hepatic, renal, or neurological disease, as determined by medical history, physical examination, laboratory tests or ECG.
18. BMI < 19 and ≥ 35 kg/m2.
19. Weight reducing drugs or appetite suppressants.
20. Estrogen replacement therapy except transdermal patch.
21. Any psychological condition which may influence the compliance with the study requirements.
22. Unstabilized antidepressant or antipsychotic medication therapy within 2 months prior to screening.
23. Subjects with a known history of alcohol abuse.
24. Subjects who received blood or plasma derivatives in the three months preceding screening.
25. Subjects who donated blood in the preceding three months of screening or intend to make a blood donation during the study, or within the three months following the study completion.
26. Subjects who have participated in another clinical study of any kind (drug or device) in the one month prior to screening.
27. Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
AE | 36 days
Laboratory values | 36 days
Vital signs | 36 days
ECG | 36 days
Patch application site reaction: Skin irritation- erythema, edema | 36 days
Patch application site reaction: Pain - Visual Analogue Scale | 36 days
Proportion of subjects (%) who discontinue the study | 36 days
Proportion of subjects (%) who discontinue the study due to AEs | 36 days
Pharmacokinetics: Somatropin exposure including Cmax, Tmax, AUC, AUC, Ke, and T1/2. | 36 days
Pharmacodynamics: Human IGF-1 levels and AUC. | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Noa Avisar, PhD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.